CLINICAL TRIAL: NCT01831362
Title: Dismantling Mindfulness: Contributions of Attention vs. Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Willoughby Britton, Assistant Professor of Psychiatry and Human Behavior, Brown University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: K23AT006328-01A1 (NIH)
Record Dates: First submitted 2013-04-10; First posted 2013-04-15 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Mild-moderate Unipolar Depression; Persistent Negative Affect
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Focused Attention (FA) (Experimental): This 8 week program consists solely of focused attention practices, i.e. selected attention to an object (breath etc) and deselection of other stimuli
  Interventions: Behavioral: Focused Attention (FA)
- Open-Monitoring (OM) (Experimental): This 8-week program consists solely of open monitoring practices, or noticing and/or labeling the contents of ongoing experience ( thoughts, body sensations, emotions, seeing, hearing etc) without focusing on or deselecting any stimuli
  Interventions: Behavioral: Open- Monitoring
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): The 8 week MBCT program follows the 2nd Edition (2012) manual (Segal, Williams, Teasdale) and includes both focused attention and open- monitoring practices
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: Focused Attention (FA)
  Arms: Focused Attention (FA)
Behavioral: Open- Monitoring
  Arms: Open-Monitoring (OM)

SUMMARY:
This study addresses NCCAM's request for research that investigates the neuropsychological mechanisms underlying mind-body therapies, and for precise criteria and better delineation of meditation practices.

The purpose of this study is to assess the clinical efficacy and mechanism of action of 2 component practices of "mindfulness meditation", i.e. focused awareness (FA) and open monitoring (OM) in comparison to each other and to the standard package, Mindfulness-Based Cognitive Therapy (MBCT).

DETAILED DESCRIPTION:
Meditation, particularly mindfulness meditation, is one of the most popular Complementary and Alternative Medicine (CAM) therapies for alleviating emotional stress, depression and anxiety. While standardized meditation-based treatment packages like Mindfulness Based Stress Reduction (MBSR) and Mindfulness-based Cognitive Therapy (MBCT) have reliably shown sustained improvements in emotional disturbances and wellbeing, they contain so many different components and practices that the active ingredient cannot be ascertained. What is commonly called "Mindfulness" meditation is actually comprised of two separate practices: 1) focused awareness practice (FA), and 2) open-monitoring practice (OM). This project aims to create separate 8 week programs for FA and OM meditations, compare their clinical efficacy and investigate their separate mechanisms of action in individuals with clinically significant levels of persistent negative affect and depression. The clinical benefit and mechanism of action of focused awareness (FA) vs open-monitoring (OM) vs MBCT will be examined with a 3-armed randomized control trial of these 8 week interventions. Outcome variables include negative affect (depression, anxiety, stress) and wellbeing. Hypothesized mediating processes include objectively measured attention, emotion regulation and the basic wakefulness on which they depend.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* ages 18-65
* mild-severe levels of depression or high level of negative affect

Exclusion Criteria:

* Current:

  * age <18 or >65
  * inability to read and write in English
  * Extremely severe levels of depression
  * active suicidal ideation
  * presence of Axis I personality disorder
  * panic disorder
  * post-traumatic stress disorder
  * obsessive-compulsive disorder
  * eating disorder, or substance abuse/dependence
  * current psychotherapy
  * change in antidepressant medication type or dosage in the last 8 weeks.

Lifetime history exclusions:

* bipolar disorder
* psychotic disorders
* persistent antisocial behavior or repeated self-harm,
* borderline personality disorder,
* organic brain damage
* regular meditation practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Inventory of Depressive Symptomatology | baseline, 8 weeks, 20 weeks
  30-item clinician administered interview about unipolar depression symptoms
change in Depression, Anxiety Stress Scale (DASS) | baseline, week 2,4,6,8, 20
  42-item self-report questionnaire on depression, anxiety and stress symptoms
change in Wellbeing Scale (WBS) | baseline, 8 weeks, 20 weeks
  73-item self-report questionnaire of psychological wellbeing

SECONDARY OUTCOMES:
Change in alpha-theta EEG power from baseline to 8 weeks | baseline and 8 weeks
  Resting/spontaneous EEG power in 5-9 Hz range
Change in Facial EMG power from baseline to 8 weeks | baseline and 8 weeks
  Facial EMG response to emotional (IAPS) photos (reactivity + regulation)
Sustained Attention to response Task (SART) | baseline, 8 weeks
  40 minuted sustained attention, go-no-go task
Difficulties in Emotion Regulation Scale (DERS) | baseline, 8 weeks, 20 weeks
  36-item self report of emotion regulation
Attention Control Questionnaire (Derryberry & Reed, 2002) | baseline, 8 weeks, 20 weeks
  20-item self report measure of attentional abilities

OTHER OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | baseline, week 3,5,7,8,20
  39-item self-report questionnaire of mindfulness skill acquisition (attention, non-reactivity)
Self-Compassion Scale (Neff 2003) | baseline, 8 weeks, 20 weeks
  26-item self report of attitudes towards oneself
Positive and Negative Affect Scale (PANAS) | week 1,2,3,4,5,6,7,8
  60-item self report of emotional states

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University Clinical and Affective Neuroscience Laboratory, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Cullen B, Eichel K, Lindahl JR, Rahrig H, Kini N, Flahive J, Britton WB. The contributions of focused attention and open monitoring in mindfulness-based cognitive therapy for affective disturbances: A 3-armed randomized dismantling trial. PLoS One. 2021 Jan 12;16(1):e0244838. doi: 10.1371/journal.pone.0244838. eCollection 2021. PMID 33434227
- [Derived] Canby NK, Eichel K, Peters SI, Rahrig H, Britton WB. Predictors of Out-of-Class Mindfulness Practice Adherence During and After a Mindfulness-Based Intervention. Psychosom Med. 2021 Jul-Aug 01;83(6):655-664. doi: 10.1097/PSY.0000000000000873. PMID 33038188
- [Derived] Britton WB, Davis JH, Loucks EB, Peterson B, Cullen BH, Reuter L, Rando A, Rahrig H, Lipsky J, Lindahl JR. Dismantling Mindfulness-Based Cognitive Therapy: Creation and validation of 8-week focused attention and open monitoring interventions within a 3-armed randomized controlled trial. Behav Res Ther. 2018 Feb;101:92-107. doi: 10.1016/j.brat.2017.09.010. Epub 2017 Sep 28. PMID 29106898
- See also: Brown University's Clinical and Affective Neuroscience Laboratory — https://www.brown.edu/research/labs/britton/